CLINICAL TRIAL: NCT03836300
Title: Piloting an Early Intervention Program for Infants With Rare Neurogenetic Disorders
Brief Title: Parent and Infant Inter(X)Action Intervention (PIXI)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Anne Wheeler, Senior Public Health Research Analyst, RTI International
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-2079
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Fragile X Syndrome; Angelman Syndrome; Prader-Willi Syndrome; Dup15Q Syndrome; Duchenne Muscular Dystrophy; Phelan-McDermid Syndrome; Rett Syndrome; Smith Magenis Syndrome; Williams Syndrome; Turner Syndrome; Klinefelter Syndrome; Chromosome 22q11.2 Deletion Syndrome; Tuberous Sclerosis; Down Syndrome
Keywords: Early intervention; Parent-Child interaction; Rare Neurogenetic Conditions; Intellectual and Developmental Disabilities
MeSH Terms: conditions — Fragile X Syndrome; Angelman Syndrome; Prader-Willi Syndrome; Muscular Dystrophy, Duchenne; Telomeric 22q13 Monosomy Syndrome; Rett Syndrome; Smith-Magenis Syndrome; Williams Syndrome; Turner Syndrome; Klinefelter Syndrome; DiGeorge Syndrome; Tuberous Sclerosis; Down Syndrome; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: The intervention, called Parent-infant Interaction Intervention (PIXI) is a comprehensive intervention provided across the first year of life for parents/caregivers of infants identified with a rare neurogenetic disorder. It includes psychoeducation around the disorder, early development, and service navigation along with parent-child interaction activities, parent coaching, and family/parent well-being support.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Infants with a rare neurogenetic condition and their parent/primary caregiver(s) (Experimental): PIXI
  Interventions: Behavioral: Parent-Infant Inter(X)action Intervention (PIXI)

INTERVENTIONS:
Behavioral: Parent-Infant Inter(X)action Intervention (PIXI) — Psychoeducation around the diagnosed disorder, early development, and service navigation along with parent-child interaction activities, parent coaching, and family/parent well-being support.

SUMMARY:
The objective is to develop and test, through an iterative process, an intervention to address and support the development of infants with a confirmed diagnosis of a neurogenetic disorder with associated developmental delays or intellectual and developmental disabilities. The proposed project will capitalize and expand upon existing empirically based interventions designed to improve outcomes for infants with suspected developmental delays.

Participants will be infants with a confirmed diagnosis of a neurogenetic disorder (e.g., fragile X, Angelman, Prader-Willi, Dup15q, Phelan-McDermid, Rhett, Smith Magenis, Williams, Turner, Kleinfelter, Down syndromes, Duchenne muscular dystrophy) within the first year of life and their parents/caregivers.

The intervention, called the Parent and Infant Inter(X)action Intervention (PIXI) is a comprehensive program inclusive of parent education about early infant development and the neurogenetic disorder for which they were diagnosed, direct parent coaching around parent-child interaction, and family/parent well-being support. The protocol includes repeated comprehensive assessments of family and child functioning, along with an examination of feasibility and acceptability of the program.

DETAILED DESCRIPTION:
The primary goal of the proposed project is to develop and test, through an iterative process, an intervention to address and support the development of infants with a rare neurogenetic condition (e.g., fragile X, Angelman, Prader-Willi, Dup15q, Phelan-McDermid, Rhett, Smith Magenis, Williams, Turner, Kleinfelter, Down syndromes, Duchenne muscular dystrophy) identified prior to emergence of symptoms. PiXI aims to utilize the foundational knowledge available around the development of and early intervention for at-risk infants to both understand the needs of and provide intervention services for families of infants diagnosed pre-symptomatically with rare neurogenetic disorders.

The investigators aim to 1) develop PIXI with a pilot sample of families, 2) test the preliminary effects of PIXI on infant and parent outcomes

ELIGIBILITY:
Inclusion Criteria:

* Infants 15 months of age or younger who have received a diagnosis which was not sought solely due to parental concerns about the infant (e.g. diagnosis due to prenatal or newborn screening, cascade testing following diagnosis of a family member).
* English must be the primary language spoken in the home because all assessment measures and intervention protocol are in English.

Exclusion Criteria:

- Infants may not be blind or have a severe hearing impairment as the intervention and assessments are not appropriate for these children.

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-11-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Social Validity and Acceptability | Completion of Phase 1 (approximately six months of age)
  A social validity measure will be completed to better understand to inquire about family satisfaction with aspects of the intervention including curriculum, timing, goals targeted, and perceived effects of the intervention.
Social Validity and Acceptability | Completion of Phase 2 (approximately twelve months of age)
  A social validity measure will be completed to better understand to inquire about family satisfaction with aspects of the intervention including curriculum, timing, goals targeted, and perceived effects of the intervention. Qualitative interviewing will be also be conducted to examine parent perceptions of feasibility and acceptability.
Fidelity | Completion of Phase 1 (approximately six months of age)
  Overall intervention fidelity will be measured by determining if the following goals were achieved:
  Enrollment target of 10-15 families 80% retention rate with at least 75% completing the 20 sessions across Phase 1 and Phase 2
Fidelity | Completion of Phase 2 (approximately twelve months of age)
  Overall intervention fidelity will be measured by determining if the following goals were achieved:
  Enrollment target of 10-15 families 80% retention rate with at least 75% completing the 20 sessions across Phase 1 and Phase 2

SECONDARY OUTCOMES:
Parent Implementation and Engagement | Across phase 1 and phase 2 engagement (approximately ages 6-months through 1-year of age)
  Internal parent implementation and engagement forms will be used to measure parent participation across both intervention phases. These components include parent readiness for the session, attention to materials, participation in topic discussion, appropriateness of intervention activity practice, and general presentation with their child.
Early Developmental Outcomes | Completion of Phase 1 (approximately 6-months of age) and completion of follow-up (approximately 36-months of age)
  Descriptive statistics around early learning, motor, communication skills, interpersonal, and adaptive skills in the sample will be derived from the Vineland Adaptive Behavior Scales, Third Edition: Parent/Caregiver Report (Vineland-3). Subdomain v-Scaled scores range from 1-24 with higher numbers indicating greater performance; while domain scores are presented in standard score formats with a range of 20-140 with higher scores indicating greater performance.
Autism Symptoms | Completion of Phase 1 (approximately 6-months of age) and completion of follow-up (approximately 36-months of age)
  A combination of measures will be used across study engagement to assess parent reported autism symptomology. These measures include the Communication and Symbolic Behavior Scale (CSBS). The parent report developmental profile is a standardized measure is completed to evaluate language and social communication predictors. A total of 57 points are available with age corresponding cutoff scores for clinical concern.
Autism Symptoms | Completion of Phase 1 (approximately 6-months of age) and completion of follow-up (approximately 36-months of age)
  A combination of measures will be used across study engagement to assess parent reported autism symptomology. These measures include the Modified Checklist for Autism in Toddlers (MCHAT). The Modified Checklist for Autism in Toddlers is a scientifically validated tool for screening children between 16 and 30 months of age that assesses risk for autism spectrum disorder (ASD).Scores range from 0-20 with corresponding ranges for cutoff scores warranting further follow-up.
Autism Symptoms | Completion of Phase 1 (approximately 6-months of age) and completion of follow-up (approximately 36-months of age)
  A combination of measures will be used across study engagement to assess parent reported autism symptomology. These measures include the Autism Diagnostic Observation Schedule, Second Edition (ADOS-2). The ADOS-2 is a semi-structured, standardized assessment of communication, social interaction, play, and restricted and repetitive behaviors. It is directly administered to the participant and behaviors are scored. Total scores range based on age of participant/module administered. Scores are calculated and compared against cutoff scores for autism spectrum and autism.
Autism Symptoms | Completion of Phase 1 (approximately 6-months of age) and completion of follow-up (approximately 36-months of age)
  A combination of measures will be used across study engagement to assess parent reported autism symptomology. These measures include the TELE-ASD-PEDS. The TELE-ASD-PEDS was developed by researchers at Vanderbilt University to assess remotely autism symptomology. The TELE-ASD-PEDS measures communication, social interaction, play, and restricted and repetitive behaviors. It is administered via telehealth and behaviors are scored. Total scores range based on age of participant/module administered. Scores are calculated and compared against cutoff scores for autism spectrum and autism.
Autism Symptoms | Completion of Phase 1 (approximately 6-months of age) and completion of follow-up (approximately 36-months of age)
  A combination of measures will be used across study engagement to assess parent reported autism symptomology. These measures include the Repetitive Behavior Scales (RBS). The RBS-EC is a questionnaire measure of restricted and repetitive behaviors designed for use in children from infancy through early school age. It is intended to capture individual differences across a broad range of behaviors associated with the repetitive behavior domain. Total scores range from 0-136 with a higher score indicating greater need/presence of behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Wheeler, PhD, Principal Investigator — RTI International
Locations (1):
- RTI International, Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No